CLINICAL TRIAL: NCT05360329
Title: Genicular Artery Embolization as Pain Treatment of Mild to Moderate Knee Osteoarthritis
Brief Title: Genicular Artery Embolization as Pain Treatment of Knee Osteoarthritis
Acronym: GETKO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Amager Hospital (Other)
Responsible Party: Principal Investigator, Louise Hindso, Doctor of Medicine, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-20081451
Record Dates: First submitted 2022-04-25; First posted 2022-05-04 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Knee Osteoarthritis
Keywords: Embolization; Geniculate Artery Embolization; Knee Osteoarthritis; Trans-arterial Embolization
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mild to moderate knee osteoarthritis (Kellgren Lawrence Score 1-3) (Experimental): Geniculate artery embolization will be performed in all eligible participants.
  Interventions: Procedure: Transarterial geniculate artery embolization

INTERVENTIONS:
Procedure: Transarterial geniculate artery embolization — The procedure will be performed in local anaesthesia. An antegrade percutaneous transfemoral approach with super-selective catheterisation of geniculate neovesselswill be performed and subsequently the target will be pruned with microspherical embolic material.

SUMMARY:
The aim of this study is to investigate the safety and efficacy of geniculate artery embolization (GAE) as pain treatment in patients with mild to moderate knee osteoarthritis.

DETAILED DESCRIPTION:
This is a single arm, prospective, pilot study investigating the safety and efficacy of GAE as pain treatment in patients with mild to moderate knee osteoarthritis. Patient related outcome measurements (PROMs), physical tests and several image modalities will be conducted.

It may form the grounding for further research in the shape of a larger randomized clinical trial.

The hypothesis is, that GAE will reduce synovitis and thereby pain in the patient group. This may secondary improve physical function and reduce consumption of analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index < 35 kg / m2.
* X-ray verified mild to moderate KOA (Kellgren Lawrence grade 1-3 [24]), obtained maximum 6 months prior to inclusion.
* Moderate to severe knee pain during walking (Visual Analog Scale (VAS) > 50 mm) - resistant to minimum 3 months physiotherapy.
* Willing, able, and mentally competent to provide informed consent.

Exclusion Criteria:

* Local infection in knee or groin areas.
* Moderate to severe pain in ipsilateral lower limb joints; VAS > 2.
* Intermittent claudication.
* Rheumatoid arthritis or seronegative arthropathies.
* Prior ipsilateral open knee surgery.
* Ipsilateral arthroscopy within 6 months.
* Ipsilateral intra-articular knee injection within 6 months.
* Current/recent (within 4 weeks) use of oral corticosteroids.
* Generalized pain syndrome (e.g. fibromyalgia) or nerve root compression syndromes.
* Pregnant or planned pregnancy during the study period.
* Lactation.
* Active malignancy.
* Known history of allergy to contrast media.
* Contra-indications for MRI (e.g. metallic foreign bodies, etc).
* Manifest hyperthyroidism.
* Diabetes (I+II).
* Liver disease.
* Only one kidney, former kidney surgery, reduced kidney function or failure (chronic or acute).
* Estimated glomerular filtration rate < 60 ml / min / 1.73 m2 (All participants: blood sample maximum 30 days prior to GAE. Participants > 60 years: another blood sample maximum 3 months prior to last MRI scan with contrast agents).
* INR > 1.4, Platelets ≤ 40 x 109 / l (All participants: blood sample maximum 30 days prior to GAE).
* Antithrombotic treatment except acetylsalicylic acid.
* Diseases affecting the bone metabolism (E.g. severe osteoporosis, Paget's disease, or hyperparathyroidism).
* American Society of Anesthesiologists classification > 3.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Changes in Visual Analog Scale (VAS) as a measure of efficacy | 6 months post GAE
  Reported as worst pain experienced during walking in the last 24 hours on a 100 mm scale from "No pain" to "Pain as bad as it could possibly be".

SECONDARY OUTCOMES:
Dexa scan | Baseline vs 6 months post GAE
  Changes in bone mineral density
Changes in Visual Analog Scale (VAS) as a measure of efficacy | 1 week, 1, 2, 3, 4, and 5 months post GAE
  Reported as worst pain experienced during walking in the last 24 hours on a 100 mm scale from "No pain" to "Pain as bad as it could possibly be".
Changes in Knee injury and Osteoarthritis Outcome Score (KOOS) | Baseline vs. 1 week, 1, 2, 3, 4, 5, and 6 months post GAE.
  KOOS assesses patient pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and knee related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms.
Changes in IPAQ (international physical activity questionnaire) | Baseline vs. 1 week, 1, 2, 3, 4, 5, and 6 months post GAE
  Questionnaire on daily physical activity
Changes in use of analgesics | Baseline vs. 1 week, 1, 2, 3, 4, 5, and 6 months post GAE
  (paracetamol, NSAID, opioid, or neuropathic agent)
Changes in 30 seconds Chair Stand Test | Baseline vs. 1 and 6 months post GAE.
  The maximum number of chair stand repetitions in a 30 second period.
Changes in Stair Climb Test | Baseline vs. 1 and 6 months post GAE.
  The time (in seconds) it takes to ascend and descend a flight of stairs.
Changes in 40 meters Fast Paced Walk Test | Baseline vs. 1 and 6 months post GAE.
  A fast-paced walking test that is timed over 4*10 meters for a total of 40 meters.
Subjective response to the treatment on a five point Likert scale | 6 months post GAE
  (none=no good at all, ineffective treatment; poor=some effect but unsatisfactory; fair=reasonable effect but could be better; good=satisfactory effect with occasional episodes of pain or stiffness; excellent=ideal response, virtually pain free)
MRI | Baseline vs. 1 and 6 months post GAE
  Changes in synovial thickness (CE-MRI), effusion (Non CE-MRI) and synovial perfusion (DCE-MRI).
Ultrasound | Baseline vs. 1 and 6 months post GAE
  Changes in synovial thickness, effusion and perfusion (doppler).

OTHER OUTCOMES:
Adverse events | 6 months
  Continually recorded from baseline till ended trial

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lönn, Professor, Study Director — Department of Radiology, University Hospital of Copenhagen, Denmark
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark